CLINICAL TRIAL: NCT04901208
Title: Acute Effects of Vaping Nicotine on Reward Processing and Inhibitory Control in Young Adults
Brief Title: Acute Effects of Vaping Nicotine on Cognition in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2000025075; 2UL1TR001863-06 (NIH); 1K01DA042937-01A1 (NIH)
Record Dates: First submitted 2021-04-30; First posted 2021-05-25 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Nicotine Addiction; Vaping
Keywords: vaping; nicotine; juul; inhibitory control; reward processing
MeSH Terms: conditions — Tobacco Use Disorder; Vaping

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Users of Juul (Active Comparator): Individuals who use Juul devices to vape nicotine
  Interventions: Drug: Nicotine pod; Drug: Placebo pod
- Controls (No Intervention): Healthy non-smokers

INTERVENTIONS:
Drug: Nicotine pod — Nicotine pods administered to individuals who use Juul
  Arms: Users of Juul
Drug: Placebo pod — Nicotine-free pods administered to individuals who use Juul
  Arms: Users of Juul

SUMMARY:
To examine reward processing and cognitive control both with and without the influence of vaporized nicotine in young adults with no history of cigarette use using EEG and fMRI. The goal is to determine whether acute nicotine administration using a Juul device would impact functional correlates of reward and inhibitory control in people who commonly use juul devices.

DETAILED DESCRIPTION:
Aim 1: To examine reward processing both with and without the influence of vaporized nicotine in young adults with no history of cigarette use using EEG and fMRI. The goal is to determine whether acute nicotine administration using a Juul device would impact functional correlates of distinguishable reward processes (anticipatory and consummatory reward) in young adults who commonly use juul devices. Predictions are that juul use will have an impact on activity in the striatum, resulting in reduced activation in fMRI and smaller amplitudes in event-related potentials (ERP) in response to reward cues and reward feedback.

Aim 2: To examine cognitive control both with and without the influence of vaporized nicotine in young adults with no history of cigarette use using EEG and fMRI. The goal is to determine whether acute nicotine administration using a Juul device would impact functional correlates of behavioral inhibition in young adults who commonly use juul devices. Predictions are that juul use will affect the inhibitory circuit, including the anterior cingulate and the dorso-lateral prefrontal cortex, resulting in decreased activation in these regions during fMRI and reductions in the FRN and P300 ERP responses in response to inhibitions and to commission errors. Predictions also include that inhibitory control behavior will be impaired after juul use.

Aim 3: To establish feasibility of naturalistic use of vaping devices for nicotine administration and observing the effects in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and to comply with all study procedures.
* For Juul users, Healthy adults between 18-30 years of age who are users of Juul (defined as reporting Juul use of 5% nicotine pods 3x per week or more and not active or previous users of cigarettes. If the first testing day reveals no cotinine in a self-reported Juul user, participants will not be permitted to continue in the study. Vaping naïve will also be defined as vaping for less than 3 months or less than 12 times. This is to prevent nicotine-naïve individuals from trying to participate for study compensation.
* Juul users will be required to already own a Juul device at screening (ie: not naive), to preclude any individuals from potentially purchasing a Juul device to join in the study. However, individuals who are 18-20 will not bring their device to the laboratory, and will instead be provided a Juul device to use.
* Controls will be healthy adults between 18-30 years of age with no history of any nicotine use. -Controls will not vape during the study at any time or have any exposure to e-cigarettes.

Exclusion Criteria:

* A serious neurological or endocrine disorder or any medical condition or treatment known to affect the brain.
* A medical condition that requires treatment with a medication with psychotropic effects.
* Occurrence of a stroke, as reported by the participant during screening.
* Any contraindications to MRI scanning (i.e., metal implants, pacemakers, etc.)
* History of loss of consciousness (LOC) for longer than 30 minutes or LOC with any neurological sequelae.
* DSM-5 criteria for intellectual disability.
* Current or a history of active neurological or psychiatric disorders, such as psychosis, bipolar illness, major depression, organic brain disease, dementia or DSM-V Axis I Psychiatric Disorder, including current alcohol or substance disorders.
* Pregnancy, as indicated by initial screening or verbal confirmation of pregnancy at one of the four testing sessions.
* (Controls only) any reports or indications (via cotinine testing) of nicotine use.
* Use of cannabis products use of CBD/THC or marijuana related products. THC testing is required at baseline and before each exposure to e-cigarettes and will exclude administration of e-cigarettes if positive. In addition, subjects who have vaped tetrahydrocannabinol (THC), cannabis (oil, dabs), or modified products with substances added that were not intended by the manufacturer, or any vaped consumables acquired from a street vendor, friend/acquaintance, or other informal source in the 90 days prior to enrollment.
* Any significant current medical condition such as neurological, cardiovascular, endocrine, renal, or hepatic pathology that would increase risk or would interfere with/mimic tobacco abstinence.
* Medical conditions increasing risk of respiratory problems in nonpatient populations: Chronic Pulmonary Conditions;
* Untreated, unresolved, acute pulmonary conditions (recurring bronchitis and Reactive airway disorder, as examples)
* Known hypersensitivity to propylene glycol.
* Planning to quit smoking with a set goal or time for quit attempt

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-04-05 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Neural correlates of reward | Activation during study session
  FMRI measures of brain activation in response to reward
Neural correlates of executive function | activation during study session
  FMRI measures of brain activation in response to tasks

CONTACTS AND LOCATIONS:
Overall Officials: Kristen P Morie, PHD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT04901208/ICF_000.pdf